CLINICAL TRIAL: NCT05110027
Title: Phase I, Open-Label, 2-Period, Single-Sequence Study to Evaluate the Mass Balance and Absorption, Disposition, Metabolism and Excretion of [14C]Enpatoran, and the Absolute Bioavailability of Enpatoran in Healthy Male Participants
Brief Title: Enpatoran Human Mass Balance and Absolute Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200569_0040; 2021-004164-10 (EudraCT Number)
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Microtracer; Microdose; Clinical Pharmacology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Enpatoran + [14C]enpatoran microtracer (Experimental)
  Interventions: Drug: Enpatoran; Drug: [14C]enpatoran microtracer
- Period 2: Enpatoran + [14C]enpatoran microdose (Experimental)
  Interventions: Drug: Enpatoran; Drug: [14C]enpatoran microdose

INTERVENTIONS:
Drug: Enpatoran — Participants will receive single oral dose of enpatoran tablet on Day 1
Drug: [14C]enpatoran microtracer — Participants will receive single oral dose of non-labeled enpatoran solution spiked with microtracer of [14C]enpatoran on Day 1 of Period 1.
  Arms: Period 1: Enpatoran + [14C]enpatoran microtracer
Drug: [14C]enpatoran microdose — Participants will receive intravenous [14C]enpatoran microdose administered at 1.5 hours after the oral dose of enpatoran on Day 1 of Period 2.
  Arms: Period 2: Enpatoran + [14C]enpatoran microdose

SUMMARY:
The purpose of Period 1 of this study is to provide a definitive quantitative characterization of the mass balance, and rates and routes of excretion of enpatoran, and to determine and quantify enpatoran and its metabolites in excreta (urine and feces) and plasma. The purpose of Period 2 of this study is to determine the absolute oral bioavailability of enpatoran. Total minimum duration of study participation for each participant is approximately 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring (blood pressure, heart rate and 12-lead electrocardiogram)
* Have a body weight within 50 to 110 kilogram (kg) and Body mass index (BMI) within the range ≥ 18.0 and ≤ 30.0 kilogram per meter square (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to Screening
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism and excretion (ADME) of drugs, or which may jeopardize the participant in case of participation in the study
* History of any malignancy
* History or presence of epilepsy, neurological disorders with seizure propensity or undiagnosed loss of consciousness, severe head trauma within 6 months or severe depression within 12 months prior to Screening), or neuropsychiatric conditions
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening, or a history of herpes zoster within 12 months prior to Screening.
* History of drug hypersensitivity ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the participant and/or outcome of the study per the Investigator's discretion
* History of alcoholism or drug abuse within 1 year prior to Screening, or evidence of such abuse as indicated by the laboratory assays conducted during Screening
* Any condition, including findings in the laboratory tests, medical history, or other Screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Period 1: Percent Urinary Recovery (feurine) of Total Radioactivity per Sampling Interval | -24-0 hours (pre-dose), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the initiation of the intravenous (IV) dose
Period 1: Percent Fecal Recovery (fefeces) of Total Radioactivity per Sampling Interval | -24-0 hours (pre-dose), 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after the initiation of the intravenous (IV) dose
Period 1: Percent Total Recovery in Urine and Feces (fetotal) of Total Radioactivity per Sampling Interval | Urine: -24-0 hours (pre-dose), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours post-dose; Feces: -24-0 hours (pre-dose), 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours post-dose of IV injection
Period 1: Pharmacokinetic Plasma and Blood Concentration of Total Radioactivity | Pre-dose (Day 1), 15, 30 minutes, 1, 1.5, 2.0, 4.0, 6.0, 8.0, 12, 24, 48, 72, 96, 120, 144, 168 hours post-dose
Period 1: Pharmacokinetic Plasma Concentration of Enpatoran | Pre-dose (Day 1), 15, 30 minutes, 1, 1.5, 2.0, 4.0, 6.0, 8.0, 12, 24, 48, 72, 96, 120, 144, 168 hours post-dose
Period 2: Pharmacokinetic Plasma and Blood Concentration of [14C]Enpatoran and Enpatoran | [14C]Enpatoran: Pre-dose, 5, 15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72 hours post-dose; Enpatoran: Pre-dose, 30 minutes, 2, 4, 6, 8, 12, 24, 48, 72 hours post-dose

SECONDARY OUTCOMES:
Period 1 and 2: Safety Profile as Assessed by Incidence of Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Laboratory Variables, Vital Signs and Electrocardiogram (ECG) Measurements | Period 1: Baseline up to Day 14; Period 2: Baseline up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https:\\bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0040
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html